CLINICAL TRIAL: NCT01177670
Title: Adiana Post-Approval Clinical Study
Brief Title: Adiana Post-Approval Clinical Study (APACS)
Acronym: APACS
Status: Terminated | Type: Observational
Why Stopped: Hologic made business decision to no longer sell or manufacture Adiana device.
Sponsor: Hologic, Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: S0210001
Record Dates: First submitted 2010-08-05; First posted 2010-08-09 (Estimated); Results first posted 2012-11-20 (Estimated); Last update posted 2012-11-20 (Estimated); Status verified 2012-10

CONDITIONS: Women Contraception
Keywords: Adiana Permanent Contraception System; women seeking permanent sterilization.

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
The Adiana Post-Approval Clinical Study (APACS) has been designed to compile information on the efficacy and safety of the Adiana Permanent Contraception System in the post market setting. Specifically, data will be collected that is relevant to the evaluation of the safety and efficacy of the Adiana System for women who desire permanent birth control by occlusion of the fallopian tubes. This study is an observational study that is not intended to test specific hypotheses.

DETAILED DESCRIPTION:
Adiana Post-Approval Clinical Study is a prospective, single armed, multi-center, observational study that is designed to provide additional efficacy and safety data regarding the FDA-approved Adiana Permanent Contraception System. This study will be conducted at 8-10 clinical sites and enroll 1000 subjects. Enrolled subjects will have baseline data collected at the time of their Adiana procedure and will then be followed for a period of 2 years with visits occurring at 3 months following the Adiana procedure, 6 months following Adiana procedure (as applicable), 12 and 24 months post relying date.

ELIGIBILITY:
Inclusion Criteria:

* Subjects who are seeking permanent sterilization
* Women 18-45 years old
* Subjects who are at risk of becoming pregnant
* Subjects willing to use alternative contraception for at least three (3) months following device placement and bilateral tubal occlusion is confirmed by HSG
* Subjects who are able to provide informed consent

Exclusion Criteria:

* Subjects who are uncertain about their desire to end fertility
* Clinical evidence of an active pelvic infection or history of a recent pelvic infection
* Has intra-uterine pathology which would prevent access to either tubal ostium or the intramural portion of either fallopian tube (i.e., large submucous fibroids, uterine adhesions, apparent uni or bilateral proximal tubal occlusion, suspected unicornuate uterus, etc.)
* Is pregnant (as evidenced by pregnancy test result) or suspects pregnancy
* Is currently less than three (3) months since her last pregnancy
* Has previously undergone a tubal ligation
* Is currently taking immunosuppressive medication (e.g., steroids)
* Has a known allergy to contrast media
* Has external pacemaker or internal cardioverter defibrillator
* Subject is unable to follow the protocol and return for follow up visits
* In the opinion of the investigator, the subject has a medical condition that precludes safe participation in the study

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Women, 18 - 45 years old, at risk for pregnancy, that are seeking permanent contraception using the Adiana Permanent Contraception System.
Sampling Method: Non-Probability Sample
Enrollment: 169 (Actual)
Dates: Start 2010-08; Study Completion 2012-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Edward Evantash, MD, Study Director — Hologic, Inc.
Locations (9):
- United States (9):
  - Sutter Medical Group, Elk Grove, California
  - WomenCare, P.C., Arlington Heights, Illinois
  - University of Missouri Health Care, Columbia, Missouri
  - Valaoras & Lewis Obstetrics and Gynecology, Winston-Salem, North Carolina
  - Complete Healthcare for Women, Columbus, Ohio
  - The Women's Center of Central Oregon, Redmond, Oregon
  - Salem Women's Clinic, Salem, Oregon
  - Western Pennsylvania Hospital, Pittsburgh, Pennsylvania
  - Ob/Gyn Associates of Danville, Danville, Virginia

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This study was designed to be conducted at 8-10 clinical sites and enroll 1000 subjects.Enrolled subjects were to have baseline data collected at the time of their procedure and then be followed for 2 years with visits occurring at 3 months following the procedure, 6 months following the procedure, 12 and 24 months post relying date.
Groups:
- Enrolled: All subjects who met enrollment inclusion/exclusion criteria, signed informed consent form, had baseline data collected and Adiana procedure performed or attempted.
Period: Overall Study
Arm/Group | Enrolled
Started | 169
Completed | 0
Not Completed | 169
Not completed — Study Terminated | 115
Not completed — Physician Decision | 50
Not completed — Withdrawal by Subject | 4

BASELINE CHARACTERISTICS:
Arm/Group | Enrolled
Number analyzed (Participants) | 169
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 169
  >=65 years | 0
Age Continuous [Mean (Standard Deviation); unit: years] | 35.8 (5.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 169
  Male | 0
Region of Enrollment [Number; unit: participants]
  United States | 169

OUTCOME MEASURES:

1. Primary Outcome: Pregnancy Rate - for Women Informed They May Rely on the Adiana System for Contraception.
Description: The primary efficacy endpoints are the one and two year pregnancy rates among women who have hysterosalpingogram (HSG)-proven bilateral occlusion and are informed that they may rely on the Adiana System for contraception.
Time Frame: At one and two years
Population: Efficacy results were not tabulated due to the early termination of the study. Only 169 of the planned 1,000 subjects (16.9%) were enrolled therefore the study is defined as incomplete, as fewer than one-third of the intended patients were enrolled.
Arm/Group | Enrolled
Number analyzed (Participants) | 0

2. Secondary Outcome: Safety Endpoints
Description: The Adiana System will be evaluated for safety on the basis of the occurrence of adverse events which are related to the study device, unanticipated or serious.
Time Frame: At one and two years
Population: Intent to treat
Measure: Number; unit: participants
Arm/Group | Enrolled
Number analyzed (Participants) | 169
participants
  Adverse Event Related to Procedure | 79
  Serious Adverse Event | 1
  Serious and Related Adverse Event | 0

ADVERSE EVENTS:
Arm/Group | Enrolled
Serious Adverse Events (participants affected / at risk) | 1/169
Other Adverse Events (participants affected / at risk) | 80/169
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Enrolled (N=169)
Hepatitis C (Infections and infestations) | 1 (1) — The serious adverse event was a diagnosis of hepatitis C that was moderate in severity, not related to the device, required outpatient treatment, and was ongoing at the termination of the study.
OTHER ADVERSE EVENTS (reported when occurring in more than 2% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Enrolled (N=169)
Pain or Cramping (General disorders) | 56 — 56: abdominal cramping, abdominal pain, cramping, left lower quadrant pain, moderate pain, pelvic cramping, pelvic cramps, pelvic pain, pelvic pain and strain, post op abdominal pain, post op pain and/or post procedure-mild pelvic pain
Bleeding (Vascular disorders) | 33 — There were 33 subjects experiencing bleeding-related adverse events (abnormal vaginal bleeding, light bleeding, moderate bleeding, scant bleeding, scant blood, scant vaginal bleeding, spotting, and/or vaginal bleeding).
Pregnancy (Reproductive system and breast disorders) | 5 — 5 subjects reporting pregnancy. 1 occurred prior to confirmation the subject could rely on Adiana.
Nausea (Gastrointestinal disorders) | 4 — 4 subjects reporting nausea (nausea and post op nausea)

LIMITATIONS AND CAVEATS:
After determining Adiana was not financially viable and would not become so, Hologic decided to discontinue manufacturing & sales. Hologic decided to terminate the study. All subjects were notified of termination and withdrawn by April 30, 2012.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less